CLINICAL TRIAL: NCT01876082
Title: PAZOPANIB Efficacy and Tolerance in Desmoids Tumors : Phase 2 Clinical Trial
Brief Title: PAZOPANIB Efficacy and Tolerance in Desmoids Tumors
Acronym: DESMOPAZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IB2011-03
Record Dates: First submitted 2012-11-06; First posted 2013-06-12 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2021-02

CONDITIONS: Progressive Desmoids Tumors
Keywords: Desmoids tumors; Pazopanib; Phase 2 clinical trial; Cross over
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAZOPANIB (Experimental): Pazopanib
  * 800 mg per day
  * oral administration
  * at least 1 hour before or 2 hours after a meal,
  * until disease progression or for 12 months maximum
  Interventions: Drug: PAZOPANIB treatment
- Vinblastine and Methotrexate (Active Comparator): vinblastine 5 mg / m², methotrexate 30 mg / m (J1, J8, J15, J21, 6 months and then J1, J15) 28 days per cycle until disease progression or for 12 months.
  Interventions: Drug: Active Comparator: Vinblastine and Methotrexate

INTERVENTIONS:
Drug: PAZOPANIB treatment — Pazopanib
  * 800 mg per day
  * oral administration
  * at least 1 hour before or 2 hours after a meal,
  * until disease progression or for 12 months maximum
  Arms: PAZOPANIB
Drug: Active Comparator: Vinblastine and Methotrexate — Active Comparator: Vinblastine and Methotrexate vinblastine 5 mg / m², methotrexate 30 mg / m (J1, J8, J15, J21, 6 months and then J1, J15) 28 days per cycle until disease progression or for 12 months.
  Arms: Vinblastine and Methotrexate

SUMMARY:
Desmoids tumors are benign soft tissues tumors characterized by aggressiveness and potential local recurrence. There is a female predominance with a sex ratio of 2/1 and median age at diagnosis is about 30 years.

Only a complete surgical excision is recommended in desmoids tumors. Some forms of desmoid tumors are recurrent and/or symptomatic and are not accessible to a conservative surgical treatment. In these clinical situations, only a medical treatment may achieve tumor control and quality of life maintenance. Place of systemic treatments in the management of desmoids tumors is poorly evaluated. Regarding chemotherapy, methotrexate and vinblastine protocol is actually the best evaluated combination, which allowed observing objective response rate between 40 and 75%. Toxicity was mainly marked by the risk of haematological toxicity.

Pazopanib is an inhibitor of multi-target tyrosine kinase, in oral form, with selective type receptors -1, -2 and -3 of VEGF receptors on the PDGFA and B, and c-Kit. It is currently under clinical development in humans in the treatment of several tumor types.

DETAILED DESCRIPTION:
This is a Phase II, randomized, multicenter, open label trial, evaluating efficacy and safety of pazopanib versus a chemotherapy protocol combining methotrexate and vinblastine in progressive and symptomatic desmoid tumors.

This study will include 72 patients in 15 centers of the French Sarcoma Group.

Patients will be treated according to therapeutic strategy allocated by randomization until documented RECIST progression and for a maximum of 12 months :

* Arm A = experimental strategy: daily oral administration of pazopanib.
* Arm B = reference strategy: methotrexate-vinblastine.

In case of documented radiological progression (RECIST criteria):

* Patients initially included in arm A will have the opportunity, as determined by the investigator, to receive arm B treatment, or leave the study,
* Patients initially included in arm B will have the opportunity, as determined by the investigator, to receive arm A treatment, or leave the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent;
2. Age ≥ 18 years;
3. ECOG ≤ 1;
4. Histologically confirmed desmoid tumor;
5. Disease progression before the patient's inclusion : completion of two similar imaging obtained within 6 months apart (a tolerance of 6 weeks is accepted)
6. Measurable target lesion (RECIST criteria) ;
7. Left ventricular ejection fraction (MUGA or ECHO) within the normal;
8. Normal hematological, renal and liver functions :

   1. Hemoglobin ≥ 9 g / dl; neutrophils ≥ 1.5 x 109 / l; platelets ≥ 100 x 109 / l; prothrombin time or INR1 ≤ 1.2 ULN or activated partial thromboplastin time ≤ 1.2 ULN;
   2. Amino alanine transferase and aspartate amino transferase ≤ 2.5 ULN;
   3. Total bilirubin ≤ 1.5 ULN;
   4. Creatinine ≤ 1.5 mg/dl or, if creatinine> 1.5 mg/dl, Creatinine clearance ≥ 50 m/min;
   5. Urinary protein / urinary creatinine (Pu / Cu) <1. If PU/Cu ≥ 1, patients must have a proteinuria below 1g/24 h
9. Women are eligible provided they:

   1. Physiologically incapable of childbearing (hysterectomy, oophorectomy, bilateral tubal ligation, menopause).
   2. Of childbearing age if they have had a negative pregnancy test in the week before the first dose of treatment.
   3. Women of childbearing potential and men must agree to take an adequate method of contraception. Permitted contraceptive methods : IUD with a documented failure rate of 1% per year, Partner's vasectomy, complete sex abstinence (for 14 days before inclusion, the test period and after cessation of treatment according to the chemotherapy as described below), dual contraception, oral contraceptives.

   Effective contraception must be implemented:
   * Up to 6 months after treatment with vinblastine
   * Up to 5 months after treatment with Methotrexate for men and up to 3 months after treatment with Methotrexate for women
   * For the duration of treatment with Pazopanib;
10. Affiliated to a social security system

Exclusion Criteria:

1. Personal history of malignancy except:

   1. Cervical intraepithelial neoplasia;
   2. Skin basal cell carcinoma;
   3. Treated localized prostate carcinoma with PSA <1;
   4. Neoplasia treated with curative intent, in remission for at least five years and considered at low risk of relapse.
2. Pretreatement by Pazopanib or Methotrexate - vinblastine;
3. Known allergy to Pazopanib, Methotrexate or vinblastine;
4. Histological sampling not available for review or biological study;
5. Clinical abnormalities which may increase the risk of gastric bleeding (not exhaustive list);

   1. Gastric tumor with known risk of bleeding;
   2. Inflammatory bowel disease or other gastrointestinal disease may increase the risk of gastric perforation.
6. Pathologies that can lead to impaired intestinal absorption (not exhaustive):

   1. Malabsorption;
   2. Major resection of small intestine or stomach.
7. Active uncontrolled infectious disease;
8. Corrected QT interval> 480 ms;
9. History of cardiovascular disease in the last 6 months:

   1. Cardiac angioplasty;
   2. Myocardial infarction;
   3. Unstable angina;
   4. Bypass surgery;
   5. Symptomatic arterial disease.
10. Congestive heart failure grade II, III or IV according to the New York Hearth Association (NYHA) classification;
11. Uncontrolled arterial hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
12. History of stroke or transient ischemic attack, pulmonary embolism or deep vein thrombosis not treated, within 6 months;
13. History of major surgery or trauma within 28 days prior the first day of treatment, or presence of a wound, fracture or non-healed ulcer;
14. Evidence of active bleeding or bleeding tendency;
15. Known endobronchial lesions and / or infiltrative lesions of the large vessels lung;
16. History of hemoptysis of more than 2.5 ml in the eight weeks preceding the first day of chemotherapy;
17. Pulmonary dysfunction, asthma, emphysema, chronic obstructive pulmonary bronchitis, pneumonia, pneumothorax, pulmonary contusion, hemothorax, distress acute respiratory syndrome, pulmonary fibrosis;
18. Severe renal dysfunction;
19. Severe hepatic dysfunction;
20. History of psoriasis, rheumatoid arthritis, alcoholism, illness or chronic liver dysfunction;
21. Any pre-existing severe or unstable medical or psychiatric condition, or other condition that may interfere with patient safety, the collection of its informed consent or adherence to treatment;
22. Patient who refused or could not stop taking banned drugs for at least 14 days (or 5 half-lives of the drug) before the first day of start of chemotherapy and for the duration of the study;
23. During cancer treatment:

    1. Radiotherapy, surgery or tumor embolization within 14 days before the 1st dose of pazobanib (arm A) or chemotherapy methotrexate, vinblastine (arm B);
    2. Chemotherapy, immunotherapy, biological treatment, experimental or hormone therapy within 14 days or 5 half-lives of medication before the first day of the pazopanib (arm A) or chemotherapy with methotrexate, vinblastine (arm B).
24. History of cancer treatment toxicity> grade 1 and / or whose the intensity increases, outside of alopecia.
25. Pregnancy and lactation
26. Concomitant treatment which can't be interrupted or replaced and which is not indicated with methotrexate:

    1. Probenecid (alone or associated with sulfamethoxazole),
    2. Trimethoprim,
    3. Acetylsalicylic acid (for methotrexate doses above 20 mg per week with the acetylsalicylic acid and used at doses analgesics or antipyretics (≥ 500 mg per dose and/or <3 g per day)or anti-inflammatory (≥ 1 g per dose and / or > 3 g per day),
    4. Phenylbutazone,
    5. Yellow fever vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09-18 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ITALIANO Antoine, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

REFERENCES:
- [Background] Toulmonde M, Pulido M, Ray-Coquard I, Andre T, Isambert N, Chevreau C, Penel N, Bompas E, Saada E, Bertucci F, Lebbe C, Le Cesne A, Soulie P, Piperno-Neumann S, Sweet S, Cecchi F, Hembrough T, Bellera C, Kind M, Crombe A, Lucchesi C, Le Loarer F, Blay JY, Italiano A. Pazopanib or methotrexate-vinblastine combination chemotherapy in adult patients with progressive desmoid tumours (DESMOPAZ): a non-comparative, randomised, open-label, multicentre, phase 2 study. Lancet Oncol. 2019 Sep;20(9):1263-1272. doi: 10.1016/S1470-2045(19)30276-1. Epub 2019 Jul 19. PMID 31331699

RESULTS

PARTICIPANT FLOW:
Groups:
- PAZOPANIB: Pazopanib
  * 800 mg per day
  * oral administration
  * at least 1 hour before or 2 hours after a meal,
  * until disease progression or for 12 months maximum
  PAZOPANIB treatment: Pazopanib
  * 800 mg per day
  * oral administration
  * at least 1 hour before or 2 hours after a meal,
  * until disease progression or for 12 months maximum
Period: Overall Study
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate
Started | 48 | 24
Safety Population (subjects having received at least one administration of treatment allocated by randomization.) | 48 | 22 (2 patients did not start control treatment)
Completed (Subjects contributing data to the primary endpoint analysis (6-month non-progression) are considered to have completed the study.) | 46 | 20
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — treatment interruption of more than 21 consecutive days observed in cycle 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate | Total
Number analyzed (Participants) | 48 | 24 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.5 [30.6 to 56.0] | 42.5 [30.5 to 54.0] | 39.8 [30.6 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 15 | 46
  Male | 17 | 9 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 48 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Remaining Alive and Progression-free at 6 Months as Per RECIST 1.1 After the Day of Randomisation (6-month Non-progression Rate).
Description: Percentage of patients remaining alive and progression-free at 6 months as per RECIST 1.1 after the day of randomisation.
  Progression is defined using New Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), or a unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: 6 months
Population: Population evaluable for efficacy included all patients who met eligibility criteria and had received at least one complete cycle or two incomplete cycles of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate
Number analyzed (Participants) | 46 | 20
percentage of participants | 84.8 [71.1 to 93.7] | 45.0 [23.1 to 68.5]

2. Secondary Outcome: Percentage of Patients Remaining Alive With Best Overall Response as Per RECIST v1.1.
Description: Best overall response is defined as the best response across all time points (RECIST v1.1). The best overall response is determined once all the data for the participant is known.
  Each patient has been assigned one of the following categories (RECIST 1.1): complete response (disappearance of all target lesions); partial response (>=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters); progression (20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) and stable disease (nor CR, PR or progression).
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate
Number analyzed (Participants) | 46 | 20
percentage of participants
  Complete response | 0 [0 to 0] | 0 [0 to 0]
  Partial response | 41.3 [27.0 to 56.8] | 30.0 [11.9 to 54.3]
  Stable disease | 54.4 [39.0 to 69.1] | 45.0 [23.1 to 68.5]
  Progression | 4.4 [0.5 to 14.8] | 20.0 [5.7 to 43.7]
  Inevaluable for response | 0 [0 to 0] | 5.0 [0.1 to 24.9]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) defined as the time from randomization to the first documented progression (as per RECIST v1.1) or death (due to any cause), whichever occurs first. Patients alive and progression free were censored at the date of last follow-up, death, or last patient contact. Progression is assessed as per RECIST v1.1. Progression-free survival is estimated as a function of time using Kaplan-Meier method.
  1- and 2-year PFS rates were reported.
Time Frame: Randomization to disease progression, or death due to any cause, whichever occurs first; until 2 years after the last patient randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate
Number analyzed (Participants) | 46 | 20
percentage of participants
  PFS rate at 1 year | 84.8 [70.7 to 92.4] | 68.6 [43.0 to 84.5]
  PFS rate at 2 years | 65.2 [49.6 to 77.0] | 68.6 [43.0 to 84.5]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) defined as the time from randomization to death (due to any cause). Patients alive were censored at the date of last follow-up or last patient contact. Overall survival was estimated as a function of time using Kaplan-Meier method.1- and 2-Year OS rates were reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate
Number analyzed (Participants) | 46 | 20
Percentage of participants
  OS rate at 1 year | 100.0 [NA to NA] — Only 1 patient from arm A died after 1 year hence insufficient patient with event to calculate the confidence limits for the 1-year OS rate. | 100.0 [NA to NA] — Only 1 patient from arm A died after 1 year hence insufficient patient with event to calculate the confidence limits for the 1-year OS rate.
  OS rate at 2 years | 97.8 [85.6 to 99.7] | 100.0 [NA to NA] — Only 1 patient from arm A died after 1 year hence insufficient patient with event to calculate the confidence limits for the 2-year OS rate.

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | PAZOPANIB | Vinblastine and Methotrexate
All-Cause Mortality (participants affected / at risk) | 1/48 | 0/22
Serious Adverse Events (participants affected / at risk) | 20/48 | 10/22
Other Adverse Events (participants affected / at risk) | 48/48 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAZOPANIB (N=48) | Vinblastine and Methotrexate (N=22)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAZOPANIB (N=48) | Vinblastine and Methotrexate (N=22)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 5 (7)
Hypothyroidism (Endocrine disorders) | 12 (13) | 0 (0)
Eye disorders - Other, specify (Endocrine disorders) | 7 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 16 (29) | 6 (6)
Bloating (Gastrointestinal disorders) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 12 (15)
Diarrhea (Gastrointestinal disorders) | 37 (60) | 9 (10)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 9 (12) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 8 (9) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (17) | 7 (11)
Nausea (Gastrointestinal disorders) | 26 (34) | 16 (19)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (3)
Vomiting (Gastrointestinal disorders) | 15 (24) | 6 (6)
Edema limbs (General disorders) | 3 (3) | 1 (2)
Fatigue (General disorders) | 40 (45) | 15 (19)
Fever (General disorders) | 3 (4) | 2 (2)
Flu like symptoms (General disorders) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 4 (4) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 8 (9) | 1 (1)
Tooth infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 15 (16) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 12 (12) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (3) | 2 (2)
GGT increased (Investigations) | 3 (8) | 3 (3)
Investigations - Other, specify (Investigations) | 6 (8) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (5) | 10 (14)
Platelet count decreased (Investigations) | 5 (6) | 0 (0)
Weight loss (Investigations) | 5 (6) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 17 (21) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (17) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (6)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Dysesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 13 (13) | 1 (1)
Headache (Nervous system disorders) | 21 (32) | 4 (5)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2) | 6 (6)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 4 (4) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 (22) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 36 (50) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0)
Hot flashes (Vascular disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 22 (27) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT01876082/Prot_SAP_000.pdf